CLINICAL TRIAL: NCT02384577
Title: Multicenter, Open-label, Non-interventional Study (NIS) to Evaluate Patient's Satisfaction and Preference, the Usability of DuoResp® SPIROMAX® and the Impact on Clinical Effects, in the Daily Routine of Asthma and COPD Treatment
Brief Title: Study to Evaluate Satisfaction and Usability of DuoResp® SPIROMAX® in Asthma and COPD Treatment
Status: Completed | Type: Observational
Sponsor: Teva Pharma GmbH (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Other Study IDs: BFS-AS-40074; DRKS00006542 (Registry Identifier: German Clinical Trials Register)
Record Dates: First submitted 2015-03-04; First posted 2015-03-10 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction | interventions — Budesonide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single group prospective treatment
  Interventions: Drug: Budesonide, Formoterol Fumarate Dihydrate

INTERVENTIONS:
Drug: Budesonide, Formoterol Fumarate Dihydrate
  Other Names: DuoResp® Spiromax®

SUMMARY:
The main aim of the study is to investigate patient satisfaction in the treatment of asthma and COPD with the new device of DuoResp® Spiromax® and patient preference. Possible difficulties in the use of the device under real-life conditions in clinical practice are investigated.

DETAILED DESCRIPTION:
The study detects the instruction expense in the use of the inhaler, reasons for the choice of the medication, or a switch in treatment of asthma or COPD.

ELIGIBILITY:
Inclusion Criteria:

* male and female adult patients with clinical diagnosis of bronchial asthma or chronic obstructive pulmonary disease
* patients on regular medication with inhaled corticosteroids and long-acting beta-2-agonists in fixed-dose combination
* patients who recently changed medication to DuoResp® Spiromax or are about to do so
* capacitated person with present declaration of consent

Exclusion Criteria:

* diseases contraindicated in accordance with the summary of product characteristic
* patients who take part in interventional clinical trials parallel or during the last 4 weeks
* patient shows conditions or diseases that might disturb the monitoring according to the physician
* patients with substance misuse in their case history (drugs, alcohol) or with other factors (e.g. serious psychiatric conditions) that limit their ability to participate in the study
* insufficient German language knowledge to understand the patient education and to complete the questionnaires in a correct manner
* patients involved in the planning and construction of the study (Teva staff and employees of the centres)
* patient is incapable of giving consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult asthma or COPD-patients
Sampling Method: Non-Probability Sample
Enrollment: 4034 (Actual)
Dates: Start 2014-07; Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction and Preference Questionnaire (PASAPQ) | 12 weeks
  Satisfaction and preference of patients treated with DuoResp® Spiromax® using PASAPQ
Practicability of the device | 12 weeks
  Investigation of practicability of the device for patients using checklist inhalation errors

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (1):
- Teva Investigational Sites, Berlin, Germany